CLINICAL TRIAL: NCT03405129
Title: Project Phoenix: Pilot Intervention for Smokers Who Are Not Ready to Quit Smoking
Acronym: Phoenix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8814
Record Dates: First submitted 2017-12-22; First posted 2018-01-19 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Smoking Cessation; Motivation
Keywords: Smoking Cessation; Smartphone App; Dynamic Treatment
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Factoid Group (Active Comparator): The Factoid group will receive a smartphone app that delivers 2 factual messages per day
  Interventions: Behavioral: Factoid
- Phoenix Group (Experimental): The Phoenix group will receive a smartphone app that includes multiple components that vary based upon the participant's smoking cessation stage
  Interventions: Behavioral: Phoenix
- Phoenix + NRT Group (Experimental): The Phoenix + (Nicotine Replacement Therapy) NRT group will receive a smartphone app that is identical to the Phoenix group, with one additional feature. Participants will be able to click an "Order Nicotine Patches and Gum" button to order NRT.
  Interventions: Behavioral: Phoenix; Behavioral: NRT order button

INTERVENTIONS:
Behavioral: Phoenix — Phoenix cessation app
  Arms: Phoenix + NRT Group; Phoenix Group
Behavioral: NRT order button — Ability to order NRT through smartphone app
  Arms: Phoenix + NRT Group
Behavioral: Factoid — Factoid app
  Arms: Factoid Group

SUMMARY:
Smoking is the leading preventable cause of death and disease in the United States. Although most smokers report that they would like to quit smoking at some point in the future, only 20% are ready to quit within the next 30 days. Importantly, studies have indicated that interventions can increase motivation and/or readiness for cessation among smokers who are not yet ready to quit and these types of intervention can increase smoking cessation attempts. Smartphone apps that offer daily information about the benefits of quitting and motivational/supportive messages that aim to increase cessation self-efficacy may increase the likelihood of initiating a smoking cessation attempt. Previous research has indicated that smoking cessation smartphone applications are feasible and well-liked by smokers who are already committed to quitting smoking. However, there are no empirically supported smartphone apps that provide dynamic smoking cessation content that is automatically matched to a smoker's current readiness to quit. This type of dynamically tailored intervention could overcome many of the barriers that have hampered the widespread use of traditional empirically supported smoking cessation treatments. The current pilot study (N=150) is a 3-armed randomized controlled smoking cessation induction trial that will determine the initial utility of a novel smartphone based intervention compared with an attention control group among smokers who are not yet ready to quit. The two intervention groups (Group 1: Phoenix App Only; Group 2: Phoenix App + Nicotine Replacement Therapy [NRT]) will receive targeted smoking cessation messaging that is matched to a participant's readiness to quit, while the attention control group (i.e., Factoid) will receive messages that are not related to smoking cessation.

DETAILED DESCRIPTION:
Description of Study Visit and Follow-Up:

Screening and Baseline Assessment Visit. Individuals who complete the online screener (i.e., REDCap) and meet initial study inclusion criteria will be invited to complete the in person screener and baseline visit at the Tobacco Treatment Research Program (TTRP). Potential participants will be provided with detailed information about the study and given the opportunity to have their questions answered within a private room to ensure confidentiality. Study staff will review the consent form with interested participants, who will be screened for eligibility on-site in a private room in the clinic. Participant eligibility for the current study will not influence eligibility for treatment at the TTRP. The Rapid Estimate of Adult Literacy in Medicine-Short Form (REALM45) will be administered to ensure that all participants are able to read at > sixth grade level (i.e., required to complete EMA and self-report questionnaires). Participants will also be asked to read aloud from the Informed Consent form. Expired carbon monoxide (CO) will be measured with a Vitalograph BreathCO carbon monoxide monitor and a Bedfont iCO carbon monoxide monitor. The purpose of using both monitors is to validate the Bedfont iCO device. Participants will be questioned in person to verify the information they provided during the REDCap screening process. Race/ethnicity, sex, cigarettes smoked per day, education, and readiness to quit smoking will be used to randomize participants to the Phoenix, Phoenix + NRT, or Factoid groups using adaptive randomization software. Participants will complete the assessment portion of the baseline visit on a laptop/tablet computer; and weight, and height will be measured in a private room to ensure confidentiality.

Participants will be instructed that the app will prompt and deliver two messages per day and that they should click the "Set New Quit Date" button when/if they want to set a smoking cessation quit date. They will be informed that the app will offer smoking cessation resources after they set a quit date.

Week 26 Follow-Up Phone Call. All participants will be asked to complete a brief 10-15 minute follow-up interview over the phone. Participants will be asked about their current smoking status, their opinions about the smartphone app, and how the app could be improved for future studies.

ELIGIBILITY:
Inclusion Criteria:

1. are ≥ 18 years of age
2. demonstrate > 6th grade English literacy level
3. possess an active Android smartphone with a data plan and an operating system version 5.2 or higher
4. agree to install the study smartphone application onto their personal phone
5. agree to complete 26 weekly assessments prompted by and completed through the study smartphone application
6. score >1 and <7 on the Readiness to Quit Ladder
7. have an expired carbon monoxide (CO) level > 7 ppm suggestive of current smoking
8. currently smoke ≥ 5 cigarettes per day
9. have no contraindications for over the counter NRT (i.e., individuals with uncontrolled blood pressure, history of myocardial infarction within the past two weeks, or current pregnancy or plans to become pregnant during the study period will be excluded)

Exclusion Criteria:

1. cannot read, speak, and understand English
2. are < 18 years of age
3. plan to quit smoking within the next 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Days of smoking abstinence | 26 weeks
  Total number of days of self-reported smoking abstinence

SECONDARY OUTCOMES:
Number of days to the first smoking cessation attempt | 26 weeks
  Number of days between the date of study enrollment and the participant's self-selected smoking cessation date. Participants will set a quit date by clicking the "Set New Quit Date" button in the study smartphone application.
Medication use | 26 weeks
  Each week, participants will be prompted by the study smartphone application to answer this question: "How many days did you use smoking cessation medications in the past 7 days?" The total number of days of medication use across the 26 week study period will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oklahoma Health Sciences Center - OTRC, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Ulm C, Chen S, Fleshman B, Benson L, Kendzor DE, Frank-Pearce S, Neil JM, Vidrine D, Businelle MS, De La Torre I. Smartphone-Based Survey and Message Compliance in Adults Initially Unready to Quit Smoking: Secondary Analysis of a Randomized Controlled Trial. JMIR Form Res. 2024 Jun 7;8:e56003. doi: 10.2196/56003. PMID 38848557
- [Derived] Businelle MS, Benson L, Hebert ET, Neil J, Kendzor DE, Frank-Pearce S, Kezbers KM, Vidrine D, Gaur A. Project phoenix: Pilot randomized controlled trial of a smartphone-delivered intervention for people who are not ready to quit smoking. Drug Alcohol Depend. 2024 Jul 1;260:111351. doi: 10.1016/j.drugalcdep.2024.111351. Epub 2024 May 31. PMID 38838477